CLINICAL TRIAL: NCT02798770
Title: Reasons for Prehospital Delay in Patients With Acute Ischemic Stroke: a Prospective Cohort Study
Brief Title: Reasons for Prehospital Delay in Patients With Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Gian Marco De Marchis, MD MSc Priv. Doz., University Hospital, Basel, Switzerland
Other Study IDs: UBE-15/64
Record Dates: First submitted 2016-06-02; First posted 2016-06-14 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke Center Basel
  Interventions: Other: No Intervention Foreseen

INTERVENTIONS:
Other: No Intervention Foreseen

SUMMARY:
Ischemic stroke is the leading cause of acquired disability among adults, and one of the main causes of death. In Switzerland, the approved time window for stroke treatment with intravenous thrombolysis after symptom onset is 4.5 h. Even within the 4.5 h time-window, however, the benefit of treatment strongly decreases as time passes.

Moreover, only around 10% patients receive thrombolytic treatment, since patients with stroke arrive too late to the hospital (prehospital delay). Despite efforts to educate the community on the symptom of stroke, prehospital delay did not decrease over time, and the reasons remain incompletely understood. Prehospital delay reduces the proportion of patients with ischemic stroke treated with thrombolysis, and reduces the odds of favorable outcome among the minority treated with thrombolysis.

This prospective cohort study aims at understanding the causes of prehospital delay among patients with acute ischemic stroke. Trained study-nurses will interview, at the bedside, patients and proxies along a standardized questionnaire on prehospital delay. Avoiding modificables causes of prehospital delay may increase the thrombolysis rate and improve outcomes after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an acute ischemic stroke hospitalized in the Stroke Center of the University Hospital Basel.

Exclusion Criteria:

* Patient not able to answer the in-person, bedside questionnaire asked by a trained study Nurse.
* Patient not willing to participate to the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an acute ischemic stroke hospitalized in the Stroke Center of the University Hospital Basel.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Prehospital Delay between between Stroke Onset and Admission to the Hospital as assessed by In-Person Interview | an average of 1 hour
  Prehospital delay will be assessed by asking the Patient or witnesses how long the time interval between stroke onset and Hospital Admission is. For instance, if stroke symptoms have onset today at 3:00 PM and the Patient gets admitted today at 4:00 PM, prehospital delay is 1 hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Stroke Center University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Ready to share/pool data. The plan to make individual participant data has to be elaborated with the interested Party.

REFERENCES:
- [Derived] Fladt J, Meier N, Thilemann S, Polymeris A, Traenka C, Seiffge DJ, Sutter R, Peters N, Gensicke H, Fluckiger B, de Hoogh K, Kunzli N, Bringolf-Isler B, Bonati LH, Engelter ST, Lyrer PA, De Marchis GM. Reasons for Prehospital Delay in Acute Ischemic Stroke. J Am Heart Assoc. 2019 Oct 15;8(20):e013101. doi: 10.1161/JAHA.119.013101. Epub 2019 Oct 2. PMID 31576773